CLINICAL TRIAL: NCT06003101
Title: Effect of Platelet-Rich Plasma, Platelet-Poor Plasma, & Bone Marrow Aspirate Concentrate Application on Functional Outcomes Following Hip Arthroscopy for Acetabular Labral Pathologies: A Prospective Randomized Controlled Trial
Brief Title: Effect of PRP, PPP, & BMAC on Functional Outcomes Following Hip Arthroscopy for Acetabular Labral Pathologies
Acronym: PRP; PPP; BMAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Scott D Martin, Principal Investigator; Director, Joint Preservation Service; Director, MGH Sports Medicine Fellowship, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P001436
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Acetabular Labrum Tear; Femoro Acetabular Impingement; Chondral Defect; Bone Marrow Aspirate Concentrate
Keywords: Acetabular Labrum Tear; Femoro Acetabular Impingement; Chondral Defect; Bone Marrow Aspirate Concentrate; Chondrolabral Junction; Osteoarthritis; Hip Arthroscopy; BMAC
MeSH Terms: conditions — Femoracetabular Impingement; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone marrow aspirate concentrate (BMAC) (Experimental): Patients randomly allocated to receive BMAC will undergo hip arthroscopy and will receive PRP/PPP/BMAC application through the PI's standardized method of harvest, processing, and application.
  Interventions: Biological: Bone marrow aspirate concentrate (BMAC)
- Control (Placebo Comparator): Patients allocated to the control cohort will receive standard of care hip arthroscopy without PRP/PPP/BMAC application.
  Interventions: Procedure: Control

INTERVENTIONS:
Biological: Bone marrow aspirate concentrate (BMAC) — Bone marrow aspiration from the body of the ilium will be performed through one of the arthroscopic portals.
  Arms: Bone marrow aspirate concentrate (BMAC)
Procedure: Control — Standard of care hip arthroscopy without bone marrow aspiration will be performed in these patients.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess the effect of PRP/PPP/BMAC application on functional outcomes after hip arthroscopy to address acetabular labral pathologies. The main questions it aims to answer are:

1. Does PRP/PPP/BMAC application improve functional outcomes after hip arthroscopy to address acetabular labral pathologies?
2. Does PRP/PPP/BMAC application reduce the arthritic burden as measured by functional outcomes following hip arthroscopy to address labral pathologies with concomitant PRP/PPP/BMAC application?

DETAILED DESCRIPTION:
1. Background Surgical management of labral pathology has evolved to reflect our current understanding of mechanism of injury and resulting hip dysfunction. Correction of labral pathology presents a technical challenge, and many techniques currently exist. Initial management of labral tears included complete resection or debridement to the bony acetabular surface of the affected region. This had the advantage of acutely reducing hip pain but was later shown by seminal biomechanical studies to compromise the mechanical integrity of the hip. With the exception of cases found to have profound degenerative changes to the labral and adjacent articular cartilage, labral resection/debridement has largely been replaced by techniques that emphasize labral tissue and blood flow preservation (i.e., repair, augmentation, reconstruction) due to a growing body of evidence reporting improved functional outcomes.

   Repair techniques focus on restoring functional anatomy by re-establishing the labrum's native position and contour on the rim of the acetabulum. Similar to repairing a torn meniscus in the knee, restoring the anatomic footprint of a torn labrum will reconstitute normal joint biomechanics. Labral injuries are often seen in the setting of femoroacetabular impingement and are a common source of early symptomatology. Therefore, during labral repair, concomitant correction of bony cam lesions, pincer lesions, or both may be necessary to prevent reinjury of the labrum. Correction of cam and pincer lesions requires femoral neck osteoplasty (trimming of femoral neck) and acetabuloplasty (trimming of the bony acetabular rim), respectively.

   Articular cartilage has limited intrinsic healing capacity and pathology frequently results in gradual and progressive tissue deterioration. Moreover, many patients presenting with hip pain in the third and fourth decade of life already have osteoarthritic changes observed at the time of arthroscopy. It has been proposed that altered biomechanics of the hip resulting from a labral tear can increase the stresses through the hip causing faster progression of cartilage wear. Moreover, previous literature has illustrated the significant association between patients with moderate to severe osteoarthritis undergoing hip arthroscopy and inferior postoperative outcomes when compared to similar patients with less osteoarthritis. Thus, while there have been notable advances in acetabular labral repair techniques, there continues to be demand for an innovation that can preserve the acetabular cartilage and chondrolabral junction in order to improve outcomes in these patients.

   Recently, given the properties of the isolated components, bone marrow aspirate concentrate (BMAC) has gained attention for its theoretical potential to treat OA and slow the progression of cartilage deterioration. BMAC contains marrow elements including mesenchymal stromal cells (MSCs), platelets, red and white blood cells, and hematopoietic precursors. Bone-marrow derived platelets contain growth factors, cytokines, and chemokines, which can promote wound healing, collagen synthesis, suppression of pro-inflammatory cytokines, production of extracellular matrix, and chondrocyte proliferation. MSCs are multipotent, non-hematopoietic stromal cells with the capacity to self-renew, proliferate, and differentiate into cartilage, bone, or fat. Numerous tissue sources can be used to isolate MSC cells, including bone marrow, adipose tissue, synovial membrane, bursa, umbilical cord blood, and periosteum. Within orthopaedic procedures, bone marrow derived MSCs (BMSCs) have been reported to be an excellent source of MSCs and are often harvested from the iliac crest, distal femur, proximal humerus, and vertebrae.

   Currently, the PI has adopted the use of a combined mixture of platelet-rich plasma (PRP), platelet-poor plasma (PPP), and BMAC that are harvested, processed, and applied during arthroscopic acetabular labral repair as his standard of care when encountering mild to moderate cartilage damage, chondrolabral junction breakdown, and isolated chondral lesions/flaps. Previous studies performed by the PI have demonstrated that harvesting bone marrow aspirate from the body of the ilium is not only a safe procedure, but also provides a concentration of connective tissue progenitor cells that is comparable to other harvest sites in the body. Furthermore, harvesting bone marrow aspirate from the body of the ilium concomitantly with arthroscopic acetabular labral repair is efficient, limits the harvesting and repair of the labrum to one procedure, and limits the procedure to only one procedural site. Regarding clinical outcomes, the PI recently published a foundational study that demonstrated that augmenting the acetabular labral repair site with bone marrow aspirate concentrate harvested from the body of the ilium resulted in significantly greater functional improvements in patients with moderate osteoarthritis compared to similar patients without BMAC application. Additionally, Kucharik et al. reported that patients with full-thickness chondral flaps treated with BMAC at the time of arthroscopic labral repair, compared to microfracture, experienced significantly greater improvements in functional outcomes at 12 months follow-up. Thus, demonstrating the possible benefits and potential of BMAC application during arthroscopic labral repair in the first randomized controlled trial (RCT) is necessary.

   The investigators are proposing the initiation of RCT) to provide Level I evidence for the investigation of the effect of PRP/PPP/BMAC application during arthroscopic acetabular labral repair. The RCT will compare postoperative outcomes between subjects that do and do not receive PRP/PPP/BMAC application during hip arthroscopy for acetabular labral pathologies using current, evidence-based, standard of care techniques. The outcomes of this study have the potential to fundamentally change the practice of hip arthroscopy across the world and lead to the improvement of countless lives. From an administrative perspective, this study could also result in future insurance coverage for the PRP/PPP/BMAC harvesting/processing/application procedure - something that is unlikely to occur from retrospective studies alone. On the other hand, if this study yields evidence that BMAC does not significantly improve the functional outcomes of patients undergoing hip arthroscopy for acetabular labral repair, it will provide critical insight to prevent patients from undergoing an additional procedure that confers minimal or no benefit at an additional cost.
2. Specific Aims and Objectives Study Aim 1: To assess the effect of PRP/PPP/BMAC application on functional outcomes after hip arthroscopy to address acetabular labral pathologies.

   Hypothesis 1.1: Subjects treated with BMAC will have significantly improved patient-reported outcome measures (PROMs) at 12 months compared to baseline.

   Hypothesis 1.2: Subjects treated without BMAC will have significantly improved PROMs at 12 months compared to baseline.

   Hypothesis 1.3: Subjects treated with BMAC will have significantly greater improvements in PROMs compared to subjects who did not receive BMAC application at 12 months compared to baseline.

   Hypothesis 1.4: Hypothesis 1.1-1.3 will hold true at 24 months and beyond.

   Study Aim 2: To evaluate the effect of arthritic burden on functional outcomes following hip arthroscopy to address labral pathologies with concomitant PRP/PPP/BMAC application.

   Hypothesis 2.1: Subjects with severe osteoarthritis (Outerbridge Grade 4, graded arthroscopically) will have inferior PROMs improvements 12 months after arthroscopic treatment of labral pathology without PRP/PPP/BMAC application, as compared to similar subjects with less severe osteoarthritis (Outerbridge Grade < or equal to 3).

   Hypothesis 2.2: Subjects with severe osteoarthritis (Outerbridge Grade 4, graded arthroscopically) will have inferior PROMs improvements 12 months after arthroscopic treatment of labral pathology with PRP/PPP/BMAC application, as compared to similar subjects with less severe osteoarthritis (Outerbridge Grade < or equal to 3).

   Hypothesis. 2.3: Hypothesis 2.1-2.3 will hold true at 24 months and beyond.

   Exploratory Hypothesis: Subjects with moderate osteoarthritis (Outerbridge Grade 2-3) treated with PRP/PPP/BMAC application will have significantly greater improvements in PROMs compared to similar subjects who did not receive PRP/PPP/BMAC application.
3. General Description of Study Design Single-blind, prospective randomized controlled trial (RCT) of patients with acetabular labral pathologies undergoing hip arthroscopy comparing outcomes of subjects receiving treatment of the labrum alone versus subjects receiving treatment of the labrum with concomitant PRP/PPP/BMAC application. Regardless of treatment allocation, no alterations will be made to the PI's surgical technique, including but not limited to initial portal placement, capsular management, addressment of the labral lesions (i.e., debridement, repair, augmentation, reconstruction), or the need to perform femoral and/or acetabular osteoplasties.

Subjects with symptomatic acetabular labral pathologies and clinically indicated for surgical intervention will be appropriately consented for hip arthroscopy by the PI. The PI routinely discusses his use of PRP/PPP/BMAC application and will briefly mention that this intervention is available, if clinically indicated during the time of surgery.

Following the surgical consenting process, potential subjects will be introduced to the study by a member of the research team. Patients not interested in participating in the study may still be offered PRP/PPP/BMAC application but will be informed that the associated cost/hospital charge must be covered out-of-pocket (i.e., direct cost to patient). Patients interested and willing to participate in the study will have their surgical consents verified to include the possible application of PRP/PPP/BMAC.

Subjects will be tracked using validated patient-reported outcomes measures (PROMs - see below), along with review of the medical record for physical exam and radiographic/advanced imaging findings to track their progress throughout the study and will continue for as long as they are a patient of the PI. Study procedures will be complete when the last enrolled subject completes 20-year follow-up and completes the corresponding surveys.

Subjects will undergo the procedure under general anesthesia and will be positioned supine on a hip distraction table. Following portal placement and establishing intra-articular access, the PI will evaluate the extent of damage and tissue quality of the labrum, chondral surfaces, transition zone cartilage, and chondrolabral junction intraoperatively, under direct arthroscopic visualization.

For patients with limited damage or degenerative changes to the labrum, articular surfaces, transition zone cartilage, and chondrolabral junction, the procedure will be carried out in standard fashion (void of any study-specific intraoperative procedures/interventions) - as PRP/PPP/BMAC application is not clinically indicated in these patients. These patients that do not meet the clinical indications for PRP/PPP/BMAC application will be stratified into a tertiary cohort to serve as 'controls' (randomization will not apply to these patients), but will continue to receive subsequent surveys via REDCap to track their functional progress and outcomes.

Conversely, for patients with evidence of damage or degenerative changes to the labrum (i.e., Beck Labral Tear Classification ≥ 1), articular surfaces (i.e., Outerbridge Grade ≥ 2), transition zone cartilage (i.e., ALAD Classification ≥ 2), and/or chondrolabral junction (i.e., Beck Chondrolabral Junction Classification ≥ 1), subsequent treatment will be dependent on their treatment allocation (outlined below). Patients will be randomized into treatment arms using a computer algorithm.

* NO TREATMENT Arm: Patients will undergo hip arthroscopy for the treatment of their labral pathology.
* TREATMENT Arm: Patients randomly allocated to receive BMAC will undergo hip arthroscopy and will receive PRP/PPP/BMAC application through the PI's standardized method of harvest, processing, and application.

Notably, bone marrow aspiration from the body of the ilium will be performed through one of the arthroscopic portals. In certain situations, pending anatomical constraints, an additional arthroscopic portal may be created to safely harvest bone marrow. However, given the normal variation in the number of arthroscopy portals created, it would be unknown to the patient, thus blinded, to whether bone marrow was harvested.

Additionally, as outlined in the informed consent document, patients will be blinded to what treatment arm they are randomized to avoid confounding the results of the PROMs they complete. Regardless of research study arm, patients will be blinded to the treatment they receive during the study period.

This off-label* use of PRP/PPP/BMAC application during hip arthroscopy has been adopted to become the PI's standard of care to date. However, to date, it has not been proven to be superior to the absence of its use in clinical practice, and thus it is being investigated as a research-specific intervention in comparison to standard of care hip arthroscopy without PRP/PPP/BMAC. Upon initiation of this proposed RCT, the PI's research fund will pay for the associated costs of the PRP/PPP/BMAC procedure if subjects are enrolled and randomized into the treatment arm of this present study. Patients that wish to receive PRP/PPP/BMAC application during their hip arthroscopy (if clinically indicated intraoperatively - upon arthroscopic visualization/assessment of the labrum/chondral surfaces/chondrolabral junction), but are not amenable to randomization/study enrollment, may opt to pay for this intervention out-of-pocket (i.e., direct charge to the patient).

By agreeing to participate in this RCT, subjects will be consenting to:

* Be randomized into a treatment arm that either will or will not receive PRP/PPP/BMAC application, if clinically indicated at the time of surgery.
* Agree to be 'blinded' to their assigned treatment allocation (i.e., subjects will not be told what treatment group they were randomized to)
* Agree to complete outcome and PROM surveys prior to surgery and at regularly scheduled intervals up until 20 years postoperatively.
* Agree to be contacted via email/phone by the study team for survey distribution, follow up with questions about survey responses, and possible reminders about survey completion.

  * The PRP/PPP/BMAC application technique is in accordance with the Federal Drug Administrations' (FDA) guidelines/considerations under section 361 of the Public Health Service (PHS) Act and Title 21 Code of Federal Regulations (CFR) Part 1271 for criterion of minimal manipulation and homologous use. Thus, the difference between un-enrolled patients and enrolled study participants is the possibility (pending randomization) for of PRP/PPP/BMAC harvest, processing, and application. Outside of the study, patients may request PRP/PPP/BMAC application during hip arthroscopy with Dr. Martin. However, these patients will be responsible for the associated out-of-pocket costs of the procedure if Dr. Martin deems PRP/PPP/BMAC application to be clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age: > or equal to 18 years
* Clinically indicated for hip arthroscopy (by the study PI) to address a labral pathology
* Willingness to participate, amenable to randomization into either treatment arm of the research study, and the ability to understand & sign the informed consent document

Exclusion Criteria:

* Non-English speaking (PROM surveys are only validated in English)
* Prior same site (i.e., ipsilateral hip) surgery, including but not limited to previous hip arthroscopy, core decompression, or periacetabular osteotomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2045-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Patient Reported Outcome Measurement (PROM) to assess the patient's functional outcomes post-surgery. Range: 0-10, with 0 being no pain and 10 being the worst pain imaginable.
Modified Harris Hip Score (mHHS) | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Patient Reported Outcome Measurement (PROM) to assess the patient's functional outcomes post-surgery. Scores range from 0 (poor) to 100 (ideal).
International Hip Outcome Tool-12 (iHOT-12) | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Patient Reported Outcome Measurement (PROM) to assess the patient's functional outcomes post-surgery. The total score is calculated as a simple mean of these responses ranging from 0 to 100, with 100 representing the best possible quality-of-life score.
Non-Arthritic Hip Score (NAHS) | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Patient Reported Outcome Measurement (PROM) to assess the patient's functional outcomes post-surgery. Scores range from 0 (poor) to 100 (ideal).
Hip Outcome Score (HOS) | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Patient Reported Outcome Measurement (PROM) to assess the patient's functional outcomes post-surgery. Scores range from 0 (poor) to 100 (ideal).
Kerlan-Jobe Orthopaedic Clinic Athletic Hip Score | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Patient Reported Outcome Measurement (PROM) to assess the patient's functional outcomes post-surgery. Scores range from 0 (poor) to 100 (ideal).
Visual Analog Scale (VAS) Pain Score | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Patient Reported Outcome Measurement (PROM) to assess the patient's functional outcomes post-surgery. Range: 0-10, with 0 being no pain and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Oswestry Low Back Disability Questionnaire (aka Oswestry Disability Index, ODI) | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Validated PROM to assess low back pain. Scores range from 0 to 50, with 0 being no disability and 50 being completed disabled.
Tegner Lysholm Knee Scoring Scale | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Validated PROM to assess knee pain. . Scores range from 0 (worse disability) to 100 (less disability).
Patient-Reported Outcomes Measurement Information System-10 (PROMIS-10) | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  Designed to be a "bottom-line" assessment of a patient's health that can be used for a wide variety of diseases. The PROMIS-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
The Pittsburgh Sleep Quality Index (PSQI): | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  The PQSI is a validated and widely used 9-question survey that is broken down into 7 scored subcomponents that measure the quality and patterns of sleep. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Patient Satisfaction, Postoperative Protocol Compliance, & Subsequent Surgeries | Baseline (pre-operative), 3 months, 6 months, 12 months, and 24 months
  A ten-question survey will be used to assess patient satisfaction with their treatment, compliance with the post-operative rehabilitation program, and track subsequent surgeries on the ipsilateral hip (i.e., revision hip arthroscopy or conversion to total hip arthroplasty) and/or lumbosacral spine.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Martin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedi A, Kelly BT. Femoroacetabular impingement. J Bone Joint Surg Am. 2013 Jan 2;95(1):82-92. doi: 10.2106/JBJS.K.01219. PMID 23283377
- [Background] Kelly BT, Weiland DE, Schenker ML, Philippon MJ. Arthroscopic labral repair in the hip: surgical technique and review of the literature. Arthroscopy. 2005 Dec;21(12):1496-504. doi: 10.1016/j.arthro.2005.08.013. PMID 16376242
- [Background] McCarthy JC, Jarrett BT, Ojeifo O, Lee JA, Bragdon CR. What factors influence long-term survivorship after hip arthroscopy? Clin Orthop Relat Res. 2011 Feb;469(2):362-71. doi: 10.1007/s11999-010-1559-2. PMID 20872105
- [Background] McCarthy JC, Noble PC, Schuck MR, Wright J, Lee J. The Otto E. Aufranc Award: The role of labral lesions to development of early degenerative hip disease. Clin Orthop Relat Res. 2001 Dec;(393):25-37. doi: 10.1097/00003086-200112000-00004. PMID 11764355
- [Background] Ferguson SJ, Bryant JT, Ganz R, Ito K. The acetabular labrum seal: a poroelastic finite element model. Clin Biomech (Bristol). 2000 Jul;15(6):463-8. doi: 10.1016/s0268-0033(99)00099-6. PMID 10771126
- [Background] Ferguson SJ, Bryant JT, Ganz R, Ito K. An in vitro investigation of the acetabular labral seal in hip joint mechanics. J Biomech. 2003 Feb;36(2):171-8. doi: 10.1016/s0021-9290(02)00365-2. PMID 12547354
- [Background] Ferguson SJ, Bryant JT, Ganz R, Ito K. The influence of the acetabular labrum on hip joint cartilage consolidation: a poroelastic finite element model. J Biomech. 2000 Aug;33(8):953-60. doi: 10.1016/s0021-9290(00)00042-7. PMID 10828325
- [Background] Larson CM, Giveans MR. Arthroscopic management of femoroacetabular impingement: early outcomes measures. Arthroscopy. 2008 May;24(5):540-6. doi: 10.1016/j.arthro.2007.11.007. Epub 2008 Jan 7. PMID 18442686
- [Background] Larson CM, Dean RS, McGaver RS, Seiffert KJ, Giveans MR. Arthroscopic Debridement Versus Refixation of the Acetabular Labrum Associated With Femoroacetabular Impingement: Updated Mean 7-Year Follow-up. Am J Sports Med. 2022 Mar;50(3):731-738. doi: 10.1177/03635465211067818. Epub 2022 Jan 31. PMID 35099305
- [Background] Larson CM, Giveans MR, Stone RM. Arthroscopic debridement versus refixation of the acetabular labrum associated with femoroacetabular impingement: mean 3.5-year follow-up. Am J Sports Med. 2012 May;40(5):1015-21. doi: 10.1177/0363546511434578. Epub 2012 Feb 3. PMID 22307078
- [Background] Espinosa N, Rothenfluh DA, Beck M, Ganz R, Leunig M. Treatment of femoro-acetabular impingement: preliminary results of labral refixation. J Bone Joint Surg Am. 2006 May;88(5):925-35. doi: 10.2106/JBJS.E.00290. PMID 16651565
- [Background] Kucharik MP, Abraham PF, Nazal MR, Varady NH, Eberlin CT, Meek WM, Martin SD. Arthroscopic Acetabular Labral Repair Versus Labral Debridement: Long-term Survivorship and Functional Outcomes. Orthop J Sports Med. 2022 Jul 7;10(7):23259671221109012. doi: 10.1177/23259671221109012. eCollection 2022 Jul. PMID 35837442
- [Background] Kucharik MP, Abraham PF, Nazal MR, Varady NH, Meek WM, Martin SD. Minimum 2-Year Functional Outcomes of Patients Undergoing Capsular Autograft Hip Labral Reconstruction. Am J Sports Med. 2021 Aug;49(10):2659-2667. doi: 10.1177/03635465211026666. Epub 2021 Jul 2. PMID 34213975
- [Background] Martin SD, Kucharik MP, Abraham PF, Nazal MR, Meek WM, Varady NH. Functional Outcomes of Arthroscopic Acetabular Labral Repair with and without Bone Marrow Aspirate Concentrate. J Bone Joint Surg Am. 2022 Jan 5;104(1):4-14. doi: 10.2106/JBJS.20.01740. PMID 34648479
- [Background] Nazal MR, McCarthy MBR, Mazzocca AD, Martin SD. Connective Tissue Progenitor Analysis of Bone Marrow Aspirate Concentrate Harvested From the Body of the Ilium During Arthroscopic Acetabular Labral Repair. Arthroscopy. 2020 May;36(5):1311-1320. doi: 10.1016/j.arthro.2019.11.125. Epub 2020 Jan 17. PMID 31958539